CLINICAL TRIAL: NCT00582959
Title: Feasibility Study of Cone Beam Imaging for Radiation Therapy Treatment Verification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-037; NCI CA59017
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Radiation Treatment for Tumors
Keywords: radiology imaging; malignancy; undergoing radiation therapy
MeSH Terms: conditions — Neoplasms

ARMS (1):
- 1 (Other): Prototype, third generation EPID based portal imaging system utilizing the MV approach.
  Interventions: Other: Cone Beam Imaging

INTERVENTIONS:
Other: Cone Beam Imaging — Prototype, third generation EPID based portal imaging system utilizing the MV approach.

SUMMARY:
The purpose of this study is to test a new technology for obtaining x-ray images of your treatment fields when you are positioned on the treatment machine, to determine whether this new system is as reliable and easy to use as conventional systems.. These so-called portal images are normally taken on a weekly basis, prior to your radiation treatment. The new portal imaging system to be tested is designed to produce better quality images than are currently achievable, but with no additional dose or added treatment time.

DETAILED DESCRIPTION:
The objective of this proposal is to test the clinical practicality of a new technology; cone beam imaging, for verification of treatment set up accuracy of cancer patients receiving radiation therapy. Currently, treatment accuracy is checked via use of 2-dimensional projection x-rays taken with the megavoltage treatment beam and electronic portal imaging devices (EPID). Typically 2 orthogonal portal images are obtained to confirm patient positioning accuracy. This method of treatment verification, however, usually provides images of poor quality and lacks true 3D information, thus making it difficult for the radiation oncologist to definitively confirm treatment accuracy. New generation EPIDs are capable of obtaining higher quality images at significantly lower imaging doses. Thus, for the same total imaging dose new generation EPIDs permit acquisition of many projection images rather than just 2 or 3. The combination of more images and higher quality images should permit more definitive assessment of treatment accuracy. We propose here to test the clinical practicality and reliability of a new prototype portal imaging system.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic proof of a malignancy suitable for radiation therapy in order to be eligible for this study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Obtain multiple (1-5) 3DCBIs on patients during the course of their radiation therapy treatments using a prototype megavoltage (MV) system and determine if the prototype imaging system is reliable and practical for routine clinical portal imaging. | conclusion of the study

SECONDARY OUTCOMES:
For some patients, in addition to obtaining 1-5 MV conebeam scans, obtain 1-2 conebeam scans using a new kilovoltage conebeam imaging system | conclusion of the study
Compare the quality and utility of the MV and kV conebeam systems. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org